CLINICAL TRIAL: NCT00714051
Title: Fall Prevention Program for Older Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E4955-R
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Accidental Falls

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fall Prevention Training (Experimental): The falls prevention training group participated in four weekly training sessions on a custom-built treadmill that produced trip-simulating perturbations (movements). While harnessed overhead to prevent actual falls, the treadmill stopped or moved suddenly. The goal for the participant was to try and prevent a fall. Each week, the level of difficulty of the task was increased.
  Interventions: Behavioral: fall prevention training
- Attention Control (Active Comparator): The attention control group participated in four weekly treadmill walking sessions at a self-selected speed.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: fall prevention training — Training on a specialized treadmill that produced trip-simulating perturbations (movements.
  Arms: Fall Prevention Training
Behavioral: Attention Control — Participants walked on a treadmill at a self-selected speed once per week for four weeks.
  Arms: Attention Control

SUMMARY:
The purpose of this study is to test the effectiveness of a fall prevention program for older adults. Participants assigned to the intervention group will train weekly on a special treadmill that will simulate tripping. Patients not assigned to the tripping program will walk on a standard treadmill.

DETAILED DESCRIPTION:
The purpose of this study is to test the effectiveness of a fall prevention program for older adults. Participants assigned to the intervention group will train weekly on a special treadmill that will simulate tripping. Patients not assigned to the tripping program will walk on a standard treadmill. The training program will last for 4 weeks. Upon completion, participants will complete a test where a trip is simulated. Those assigned to the intervention group will test one additional time as well.

ELIGIBILITY:
Inclusion Criteria:

* 65-80 yr old,
* normal reflexes and muscle tone

Exclusion Criteria:

* lower extremity fracture or surgery last 5 yrs
* back surgery or disc herniation last 5 yrs
* noticeable gait impairment,
* low back pain,
* decreased disease-related vision,
* dizziness,
* history of heart problems,
* bone mineral density <.65,
* mini-mental score <24

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-10; Primary Completion 2012-02 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen G. Collins, PhD RN, Principal Investigator — Edward Hines Jr. VA Hospital
Locations (1):
- Edward Hines, Jr. VA Hospital, Hines, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the general medical clinics, nuclear medicine department and electronic medical record. Letters of invitation were sent to eligible participants. Recruitment began in January 2009 and ended in August 2011. .
Pre-assignment Details: 92 participants were screened for eligibility in the study. 55 participants were randomized and 37 were not randomized. Reasons for not being randomized are: 13 = bone mineral density of less than .65 gm/cm2; 11 =could not meet time commitments of study; 3=orthopedic problems; 10=other reasons
Groups:
- Falls Prevention Training: The falls prevention training group participated in four weekly training sessions on a custom-built treadmill that produced trip-simulating perturbations (movements). While harnessed overhead to prevent actual falls, the treadmill stopped or moved suddenly. The goal for the participant was to try and prevent a fall. Each week, the level of difficulty of the task was increased.
- Control: The control group participated in four weekly treadmill walking sessions at a self-selected speed.
Period: Overall Study
Arm/Group | Falls Prevention Training | Control
Started | 27 | 28
Completed | 26 | 27
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Falls Prevention Training Group: The falls prevention training group participated in four weekly training sessions on a custom-built treadmill that produced trip-simulating perturbations (movements). While harnessed overhead to prevent actual falls, the treadmill stopped or moved suddenly. The goal for the participant was to try and prevent a fall. Each week, the level of difficulty of the task was increased.
- Control Group: The control group participated in four weekly treadmill walking sessions at a self-selected speed.
- Total: Total of all reporting groups
Arm/Group | Falls Prevention Training Group | Control Group | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (4.2) | 70.9 (4.3) | 71.9 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 25 | 26 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 25 | 28 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 28 | 55
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55
Co-morbidities [Mean (Standard Deviation); unit: co-morbidities] | 2.6 (1.6) | 3.1 (2.2) | 2.9 (1.9)
Bone mineral density [Mean (Standard Deviation); unit: gm/cm2] | 0.94 (0.1) | 0.90 (0.11) | 0.92 (0.11)
Six minute walk [Mean (Standard Deviation); unit: meters] | 546 (90) | 545 (102) | 545 (96)
Modified Falls Efficacy Scale [Mean (Standard Deviation); unit: units on a scale] — The Modified Falls Efficacy scale measures self-perceived fear of falling during the completion of 14 common activities. A score of 0=not confident at all and a score of 10=completely confident. The items are summed to form a total score. The higher score is the better score. The range of scores is 0-140.
  units on a scale | 136.5 (9.9) | 136.3 (10.5) | 136.4 (10.1)
Sit and reach flexibility [Mean (Standard Deviation); unit: Centimeters] | 15.4 (12.8) | 16.2 (9.4) | 15.8 (11.1)
Quadriceps strength [Mean (Standard Deviation); unit: foot pounds] | 89.5 (25.6) | 89.5 (20.4) | 89.5 (22.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Fell on a Tripping Test
Description: Participants completed a tripping test upon completion of the 4 weeks training period. Participants walked along a platform while harnessed to an overhead rail. Participants walked at a self-selected pace knowing that they will be tripped but do not know how or when the trip will be induced. The trip is induced by an obstruction that deploys from the floor. A decoy rope was laid across the pathway about 3 meters before the trip to intentionally mislead the participant to expect the trip at that point. This expectation affects gait and response to a trip. The participant was tripped on the 3rd set of 10 walking trials.
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- Attention Control: The control group participated in four weekly treadmill walking sessions at a self-selected speed.
Arm/Group | Falls Prevention Training | Attention Control
Number analyzed (Participants) | 26 | 27
participants | 2 | 4
Statistical Analysis 1: Comparison: Falls Prevention Training vs Attention Control; The number of participants who fell on the tripping trial in each group were compared using Chi-square analysis; Test type: Superiority or Other; p = 0.45, Chi-squared

ADVERSE EVENTS:
Arm/Group | Falls Prevention Training | Attention Control
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/28
Other Adverse Events (participants affected / at risk) | 0/27 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Falls Prevention Training (N=27) | Attention Control (N=28)
Death (Cardiac disorders) | 0 (0) | 1 (1) — Participant was found dead at home by spouse. Cause was presumed cardiac. Participant had completed baseline testing and was randomized but had not completed any control study visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No